CLINICAL TRIAL: NCT01340144
Title: Evaluation of Patellar Crepitus Following PFC Sigma vs. PFC Sigma HP Total Knee Arthroplasty: Does Femoral Component Design Make a Difference?
Brief Title: Evaluation of Patellar Crepitus Following Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Colorado Joint Replacement (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: IIS-000112
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Results first posted 2015-03-05 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Total Knee Replacement
Keywords: total knee replacement; patellar crepitus; Replacement of knee joint

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PFC Sigma PS TKA: one group received primary TKA using the PFC Sigma PS TKA
- PFC Sigma HP PS TKA: One group received primary TKA using the PFC Sigma HP PS TKA.

SUMMARY:
Analyze clinical data for a group of subjects implanted with a new surgical device designed to reduce the incidence of patellar crepitus following PCL-substituting TKA and compare that to a control group of subjects implanted with a TKA design known to have an incidence of patellar crepitus of approximately 5%.

DETAILED DESCRIPTION:
Patellar crepitus and clunk following posterior cruciate substituting total knee arthroplasty is a persistent problem with a reported incidence as high as 14%. The development of this complication necessitates additional surgery in some patients. Numerous etiologies have been reported including design of the femoral component. Due to a higher than desired incidence of patellar crepitus with the PFC Sigma PS TKA, design modifications of the trochlear groove of the femoral component were introduced with the release of the PFC Sigma HP PS femoral component. The purpose of the proposed study is to evaluate the incidence of patellar crepitus after posterior cruciate substituting TKA utilizing the PFC Sigma vs. the PFC Sigma HP PS femoral components.

ELIGIBILITY:
Inclusion Criteria:

* subjects that received primary total knee replacement

Exclusion Criteria:

* Did not return for follow - up appointments Required any post operative manipulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colorado Joint replacement clinic
Sampling Method: Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Kim, MD, Principal Investigator — Porter Adventist Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- PFC Sigma PS TKA (Total Knee Arthroplasty): One group received primary TKA using the PFC Sigma PS TKA
- PFC Sigma HP PS TKA (Total Knee Arthroplasty): One group received primary TKA using the PFC Sigma HP PS TKA.
Period: Overall Study
Arm/Group | PFC Sigma PS TKA (Total Knee Arthroplasty) | PFC Sigma HP PS TKA (Total Knee Arthroplasty)
Started | 625 | 625
Completed | 553 | 567
Not Completed | 72 | 58

BASELINE CHARACTERISTICS:
Groups:
- PFC Sigma HP PS TKA (Total Knee Arthoplasty): One group received primary TKA using the PFC Sigma HP PS TKA.
- Total: Total of all reporting groups
Arm/Group | PFC Sigma PS TKA (Total Knee Arthroplasty) | PFC Sigma HP PS TKA (Total Knee Arthoplasty) | Total
Number analyzed (Participants) | 625 | 625 | 1250
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 65.6 [46.9 to 84.3] | 65.6 [47.3 to 83.9] | 65.6 [46.9 to 84.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 350 | 352 | 702
  Male | 275 | 273 | 548
Region of Enrollment [Number; unit: participants]
  United States | 625 | 625 | 1250

OUTCOME MEASURES:

1. Primary Outcome: Evaluate for the Incidence of Patellar Crepitus Requiring Non-operative vs. Operative Treatment of Both the Study and Control Groups at a Minimum of 12 Months Following the TKA (Total Knee Arthroplasty) Procedure in Each Subject.
Description: The incidence of patellar crepitus and clunk will be statistically compared between the study (PFC Sigma HP PS TKA) and control (PFC Sigma PS TKA groups). Based on a strength analysis to determine a theoretical reduction in the incidence of patellar crepitus from 5% to 2%, a study group of 625 subjects in both the control and study ggroups will be required. Each group will also be statistically analyzed using the following variables: overall crepitus incidence, incidence of crepitus requiring only non-operative treatment vs. those requiring operative treatment to manage this complication.
Time Frame: Two years after TKA (Total Knee Arthroplasty) procedure
Measure: Number; unit: participants
Arm/Group | PFC Sigma PS TKA (Total Knee Arthroplasty) | PFC Sigma HP PS TKA (Total Knee Arthroplasty)
Number analyzed (Participants) | 553 | 567
participants
  Positive Crepitus | 78 | 82
  Symptomatic Crepitus | 31 | 24
  Operative Crepitus | 18 | 7

ADVERSE EVENTS:
Arm/Group | PFC Sigma PS TKA (Total Knee Arthroplasty) | PFC Sigma HP PS TKA (Total Knee Arthroplasty)
Serious Adverse Events (participants affected / at risk) | 45/625 | 29/625
Other Adverse Events (participants affected / at risk) | 0/625 | 0/625
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFC Sigma PS TKA (Total Knee Arthroplasty) (N=625) | PFC Sigma HP PS TKA (Total Knee Arthroplasty) (N=625)
Failed total knee due to infection (Infections and infestations) | 4 (4) | 1 (1)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) — Colon cancer with liver metastases
Failed total knee due to arthrofibrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Failed TKA due to chronic patellofemoral and mild tibiofemoral instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 3 (3) — Unknown cause
Death (Cardiac disorders) | 1 (1) | 0 (0) — Cause of Death: MI
Periprosthetic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Cerebellar tumor, esophageal cancer
Dehiscence (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Chronic lateral patellar irritation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Bladder cancer
Death (Infections and infestations) | 1 (1) | 0 (0) — Cause of death: sepsis
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) — Lung cancer
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Lung cancer
Hemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 15 (15) | 4 (4)
Below knee amputation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Total hip replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Hip dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Femoral fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Nondisplaced femoral neck fracture
Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cause of death: Pneumonia
Death (Cardiac disorders) | 0 (0) | 4 (4)
Failed TKA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Failed TKA due to quadriceps tendon rupture
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Conralateral TKA (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Lumbar stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hetrotrophic bone formation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peroneal nerve entrapment (Nervous system disorders) | 0 (0) | 1 (1)
Achilles tendon rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No